CLINICAL TRIAL: NCT02598557
Title: Alternative Dosing of Exemestane in Postmenopausal Women With Stage 0-II ER-Positive Breast Cancer: A Randomized Presurgical Trial
Brief Title: Alternative Dosing of Exemestane Before Surgery in Treating Postmenopausal Patients With Stage 0-II Estrogen Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2015-01821; NCI-2015-01821 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HHSN26120120034I; N01-CN-2012-00034; 2016-0276 (Other: M D Anderson Cancer Center); MDA2014-04-01 (Other: DCP); N01CN00034 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Stage 0 Breast Cancer AJCC v6 and v7; Stage I Breast Cancer AJCC v7; Stage IA Breast Cancer AJCC v7; Stage IB Breast Cancer AJCC v7; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — exemestane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I: Exemestane 25 mg QD (Experimental): Patients receive exemestane PO QD on days 1-7. Cycles repeat every 7 days for 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery on days 29, 36, or 43.
  Interventions: Drug: Exemestane; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery
- Arm II: Exemestane 25 TIW (exemestane, placebo) (Experimental): Patients receive exemestane PO QD on days 1, 3, and 5. Patients also receive placebo PO QD on days 2, 4, 6, and 7. Cycles repeat every 7 days for 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery on days 29, 36, or 43.
  Interventions: Drug: Exemestane; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery
- Arm III: Exemestane 25 mg QW (exemestane, placebo) (Experimental): Patients receive exemestane PO QD on day 1 and placebo PO QD on days 2-7. Cycles repeat every 7 days for 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery on days 29, 36, or 43.
  Interventions: Drug: Exemestane; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm II: Exemestane 25 TIW (exemestane, placebo); Arm III: Exemestane 25 mg QW (exemestane, placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase IIb trial studies how well alternative dosing of exemestane before surgery works in treating in postmenopausal patients with stage 0-II estrogen positive breast cancer. Chemoprevention is the use of drugs to keep breast cancer from forming or coming back. The use of exemestane may treat early stage (stage 0-II) breast cancer. Comparing the exemestane standard dose regimen versus two alternative, less frequent dose regimens may decrease undesirable symptoms and have similar efficacy in reducing serum estradiol.

DETAILED DESCRIPTION:
We have conducted an international, multicenter, pre-surgical double-blind non-inferiority phase IIb study in which a total of 180 participants have been randomized to receive either exemestane 25 mg/day (Exemestane 25 mg QD) or 25 mg/ three times a week (Exemestane 25 mg TIW) or a single dose of 25 mg/week (Exemestane 25 mg QW) for a minimum of 4 up to 6 weeks. Participants were stratified by center and BMI (<25 kg/m2 vs >25 kg/m2).

Participants were histologically confirmed ER-positive (ER >10%) primary breast cancer patients who were candidates for breast surgery. Postmenopausal women younger than 76 years of age with cT0-2, cN0-1, Mx or women with larger tumors who refuse neo-adjuvant therapy before surgery were eligible. No previous treatment for breast cancer was allowed.

Complete physical exam and safety lab tests have been performed at baseline and at the end of treatment (28+1, 35+1, 42+1 days). Phone contact occurred on day 1 and a week before surgery (+3 days). Participants experiencing persistent adverse events (certainly, probably, and possibly treatment-related) have been monitored 20-30 days after study completion.

Biomarkers: blood samples were collected at baseline and the end of treatment (fasting blood for biomarkers collected prior to randomization and either on the day of surgery or the day before; fasting strongly recommended but not mandated), tissue samples collected from the diagnostic or research biopsy and at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (postmenopausal: age >= 60 years, or amenorrhea >= 12 months, or bilateral oophorectomy, or - in women with hysterectomy only - follicle stimulating hormone [FSH] in the menopausal levels as per local institutional guidelines if < 60 years old) with histologically-confirmed estrogen receptor (ER)-positive (>= 10%) primary breast cancer stage cT0-2, cN0-1, Mx; women with larger tumors who refuse chemotherapy (chemo) and/or endocrine neoadjuvant therapy can be eligible
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,500/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional ULN
* Serum creatinine =< 1.5 times institutional ULN
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Body mass index (BMI) < 18.5 Kg/m^2
* Previous treatment for breast cancer including chemotherapy, endocrine therapy and radiotherapy; women with prior ductal breast carcinoma in situ (DCIS) who were treated with surgery only and whose treatment ended >= 2 years prior to enrollment are eligible for the trial
* Women who are planned to receive neoadjuvant therapy
* Participants may not be receiving investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to exemestane
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Other co-existing invasive malignancies (with the exclusion of basal cell carcinoma or skin squamous cell carcinoma) diagnosed during the last 2 years before randomization
* History of severe osteoporosis (T score =< -4 either spine or hip), or presence of vertebral fracture
* Use of systemic hormone replacement therapy (HRT) in the last 30 days prior to the randomization; the use of non-systemic estrogen (such as vaginal estrogen use) is allowed
* Use of any chemopreventive agents (selective estrogen receptor modulators [SERM]) in the last 3 months
* Concomitant use of CYP3A4 inducer medication (rifampicin, phenytoin, carbamazepine, phenobarbital, and St. John's wort)

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernardo Bonanni, Principal Investigator — European Institute of Oncology
Locations (5):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas
- Italy (2):
  - Galliera Hospital, Genoa
  - European Institute of Oncology, Milan

REFERENCES:
- [Derived] Serrano D, Johansson H, Bertelsen BE, Gandini S, Mellgren G, Thomas P, Crew KD, Kumar NB, Macis D, Aristarco V, Guerrieri-Gonzaga A, Lazzeroni M, D'Amico M, Buttiron-Webber T, Briata IM, Spinaci S, Galimberti V, Vornik LA, Vilar E, Brown PH, Heckman-Stoddard BM, Szabo E, Bonanni B, DeCensi A. Drug and biomarker tissue levels in a randomized presurgical trial on exemestane alternative schedules. J Natl Cancer Inst. 2024 Dec 1;116(12):1979-1982. doi: 10.1093/jnci/djae183. PMID 39110531
- [Derived] Serrano D, Gandini S, Thomas P, Crew KD, Kumar NB, Vornik LA, Lee JJ, Veronesi P, Viale G, Guerrieri-Gonzaga A, Lazzeroni M, Johansson H, D'Amico M, Guasone F, Spinaci S, Bertelsen BE, Mellgren G, Bedrosian I, Weber D, Castile T, Dimond E, Heckman-Stoddard BM, Szabo E, Brown PH, DeCensi A, Bonanni B. Efficacy of Alternative Dose Regimens of Exemestane in Postmenopausal Women With Stage 0 to II Estrogen Receptor-Positive Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2023 May 1;9(5):664-672. doi: 10.1001/jamaoncol.2023.0089. PMID 36951827
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 participants were not randomized (25 not eligible, 20 withdrew consent, 5 other reasons)
Groups:
- Exemestane 25 mg QD: 1 tablet of exemestane 25 mg a day for up to 6 weeks
- Exemestane 25 mg TIW: 1 tablet of exemestane 25 mg a day (on days 1, 3, 5) and 1 tablet of placebo on days 2, 4, 6, 7 for up to 6 weeks
- Exemestane 25 mg QW: 1 tablet of exemestane 25 mg a day (on day 1) and 1 tablet of placebo on days 2 to 7 for up to 6 weeks
Period: Overall Study
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Started | 59 | 58 | 63
Completed | 55 | 56 | 60
Not Completed | 4 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Participant did not start treatment | 2 | 1 | 1
Not completed — Unavailable specimen for endpoint evaluations | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW | Total
Number analyzed (Participants) | 57 | 57 | 62 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 32 | 29 | 86
  >=65 years | 32 | 25 | 33 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [60 to 71] | 63 [60 to 69] | 65 [61 to 70] | 64 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 62 | 176
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10 | 20
  Not Hispanic or Latino | 52 | 49 | 51 | 152
  Unknown or Not Reported | 2 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 8
  White | 49 | 51 | 55 | 155
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 3 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 28 | 31 | 34 | 93
  Italy | 29 | 26 | 28 | 83
Circulating levels of unconjugated estradiol SPE (Solid phase extraction) [Median (Inter-Quartile Range); unit: pmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  pmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 21.6 [12.0 to 35.6] | 22.4 [12.7 to 33.4] | 20.6 [13.6 to 31.5] | 21.3 [12.5 to 32.8]
Circulating levels of unconjugated estradiol LLE (Liquid liquid extraction) [Median (Inter-Quartile Range); unit: pmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  pmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 21.2 [13.5 to 34.1] | 20.9 [12.6 to 32.5] | 19.7 [11.9 to 28.9] | 20.5 [12.4 to 33.8]
Circulating levels of unconjugated estrone SPE(Solid phase extraction) [Median (Inter-Quartile Range); unit: pmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  pmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 104.3 [73.8 to 141.0] | 99.4 [69.4 to 137.6] | 92.2 [66.7 to 122.8] | 98.7 [70.0 to 132.5]
Circulating levels of unconjugated estrone LLE (Liquid liquid extraction) [Median (Inter-Quartile Range); unit: pmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  pmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 101.0 [69.6 to 143.0] | 96.2 [72.1 to 147.5] | 93.4 [69.5 to 132.0] | 98.3 [70.2 to 137.0]
Circulating levels of total estrone [Median (Inter-Quartile Range); unit: pmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  pmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 294.7 [182.6 to 451.4] | 302.2 [160.0 to 429.9] | 246.1 [164.0 to 362.1] | 279.9 [169.9 to 419.2]
Circulating levels of estrone sulfate [Median (Inter-Quartile Range); unit: pmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  pmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 581.9 [363.6 to 918.9] | 625.8 [324.7 to 955.6] | 452.3 [315.1 to 710.6] | 560.4 [330.8 to 853.4]
Circulating levels of androstenedione [Median (Inter-Quartile Range); unit: nmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  nmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 1.5 [1.0 to 1.9] | 1.7 [1.1 to 2.5] | 1.4 [1.1 to 2.0] | 1.5 [1.1 to 2.0]
Circulating levels of testosterone [Median (Inter-Quartile Range); unit: nmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  nmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 0.6 [0.4 to 0.9] | 0.7 [0.4 to 1.1] | 0.6 [0.4 to 0.9] | 0.6 [0.4 to 0.9]
Circulating levels of testosterone CLIA (Chemiluminescent immunoassay) [Median (Inter-Quartile Range); unit: nmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  nmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 0.447 [0.259 to 0.853] | 0.512 [0.331 to 0.860] | 0.425 [0.238 to 0.702] | 0.477 [0.284 to 0.797]
Circulating levels of SHBG (Sex Hormone-Binding Globulin) [Median (Inter-Quartile Range); unit: nmol/L] — Population: The numbers are lower because there were no specimen available for analysis.
  nmol/L
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 53.4 [39.1 to 64.0] | 47.9 [36.6 to 65.1] | 50.1 [31.9 to 67.8] | 50.6 [35.6 to 65.5]
Circulating levels of total cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Population: The numbers are lower because there were no specimen available for analysis.
  mg/dL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 205 [181 to 233] | 208 [182 to 226] | 220 [202 to 247] | 213 [188 to 240]
Circulating levels of High density lipoprotein (HDL) cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Population: The numbers are lower because there were no specimen available for analysis.
  mg/dL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 62 [55 to 72] | 59 [48 to 71] | 57 [50 to 67] | 59 [51 to 69]
Circulating levels of Low density lipoprotein (LDL) cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Population: The numbers are lower because there were no specimen available for analysis.
  mg/dL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 122.7 [95 to 145.6] | 120.4 [101.2 to 147.6] | 132.3 [110.4 to 162.8] | 123.6 [103.6 to 151.8]
Circulating levels of triglycerides [Median (Inter-Quartile Range); unit: mg/dL] — Population: The numbers are lower because there were no specimen available for analysis.
  mg/dL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 104 [89 to 142] | 92 [75 to 151] | 119 [94 to 169] | 108 [81 to 148]
Circulating levels of insulin [Median (Inter-Quartile Range); unit: uU/mL] — Population: The numbers are lower because there were no specimen available for analysis.
  uU/mL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 7.6 [5.8 to 10.6] | 8.1 [5.8 to 12.4] | 7.9 [5.3 to 12.9] | 8.0 [5.7 to 11.5]
Baseline levels of serum glucose [Median (Inter-Quartile Range); unit: mg/dL] — Population: The numbers are lower because there were no specimen available for analysis.
  mg/dL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 96 [89 to 103] | 98 [92 to 110] | 95 [90 to 105] | 97 [90 to 106]
HOMA IR [Median (Inter-Quartile Range); unit: HOMA IR Index] — Insulin Resistance Index (HOMA-IR) measures insulin resistance, calculated by fasting insulin (mU/L) multiplied by fasting glucose (mmol/L), and divided by a constant (22.5). A higher score indicates higher insulin resistance. Population: The numbers are lower because there were no specimen available for analysis.
  HOMA IR Index
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 1.76 [1.34 to 2.61] | 1.99 [1.49 to 3.25] | 1.96 [1.32 to 3.15] | 1.94 [1.35 to 2.90]
Circulating levels of adiponectin [Median (Inter-Quartile Range); unit: µg/mL] — Population: The numbers are lower because there were no specimen available for analysis.
  µg/mL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 10.99 [7.84 to 14.21] | 8.82 [6.54 to 11.66] | 8.99 [6.56 to 12.92] | 9.5 [6.81 to 13.28]
Circulating levels of leptin [Median (Inter-Quartile Range); unit: ng/mL] — Population: The numbers are lower because there were no specimen available for analysis.
  ng/mL
    number analyzed (Participants) | 55 | 56 | 60 | 171
    (all) | 35.1 [23.9 to 75.8] | 41.7 [18.7 to 65.1] | 38.5 [22.5 to 72.1] | 36.6 [20.6 to 69.3]
Tissue biopsy estrogen receptor level (centralized evaluation) [Median (Inter-Quartile Range); unit: Percentage of positive tumor cells] — Population: The numbers are lower because there were no specimen available for analysis.
  Percentage of positive tumor cells
    number analyzed (Participants) | 52 | 53 | 55 | 160
    (all) | 99 [95 to 99] | 99 [97 to 99] | 99 [95 to 99] | 99 [95 to 99]
Tissue biopsy progesteron receptor level (centralized evaluation) [Median (Inter-Quartile Range); unit: Percentage of positive tumor cells] — Population: The numbers are lower because there were no specimen available for analysis.
  Percentage of positive tumor cells
    number analyzed (Participants) | 52 | 53 | 55 | 160
    (all) | 65 [10 to 95] | 70 [10 to 99] | 70 [8 to 95] | 70 [10 to 95]
Tissue biopsy Ki-67 cancer tissue (centralized evaluation) [Mean (Inter-Quartile Range); unit: Percentage of positive tumor cells] — Population: The numbers are lower because there were no specimen available for analysis.
  Percentage of positive tumor cells
    number analyzed (Participants) | 52 | 53 | 55 | 160
    (all) | 13 [7 to 17] | 13 [7 to 20] | 12 [6 to 19] | 12 [7 to 18]
Tissue biopsy Ki-67 adjacent non cancer tissue (centralized evaluation) [Median (Inter-Quartile Range); unit: Percentage of positive tumor cells] — Population: The numbers are lower because there were no specimen available for analysis.
  Percentage of positive tumor cells
    number analyzed (Participants) | 28 | 22 | 27 | 77
    (all) | 1 [1 to 2] | 1 [0 to 3] | 1 [1 to 2] | 1 [1 to 2]
UGT2B17 Copy number variation distribution by arm [Number; unit: count] — Population: The numbers are lower because there were no specimen available for analysis.
  count
    2: number analyzed (Participants) | 53 | 54 | 57 | 164
    2 | 22 | 23 | 19 | 64
    1: number analyzed (Participants) | 53 | 54 | 57 | 164
    1 | 22 | 26 | 30 | 78
    0: number analyzed (Participants) | 53 | 54 | 57 | 164
    0 | 9 | 5 | 8 | 22
CYP19A1 rs10046 distribution by arm [Count of Participants; unit: Participants] — Population: The numbers are lower because there were no specimen available for analysis.
  Participants
    wt/wt: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/wt | 11 | 15 | 12 | 38
    wt/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/v | 31 | 31 | 33 | 95
    v/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    v/v | 11 | 8 | 12 | 31
CYP19A1 rs4646 distribution by arm [Count of Participants; unit: Participants] — Population: The numbers are lower because there were no specimen available for analysis.
  Participants
    wt/wt: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/wt | 29 | 25 | 35 | 89
    wt/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/v | 18 | 25 | 17 | 60
    v/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    v/v | 6 | 4 | 5 | 15
CYP3A4*22 rs35599367 distribution by arm [Count of Participants; unit: Participants] — Population: The numbers are lower because there were no specimen available for analysis.
  Participants
    wt/wt: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/wt | 49 | 51 | 56 | 156
    wt/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/v | 4 | 3 | 1 | 8
    v/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    v/v | 0 | 0 | 0 | 0
SLCO1B1 rs4149056 distribution by arm [Count of Participants; unit: Participants] — Population: The numbers are lower because there were no specimen available for analysis.
  Participants
    wt/wt: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/wt | 37 | 38 | 41 | 116
    wt/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/v | 13 | 13 | 16 | 42
    v/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    v/v | 3 | 3 | 0 | 6
SLCO1B1 rs10841753 distribution by arm [Count of Participants; unit: Participants] — Population: The numbers are lower because there were no specimen available for analysis.
  Participants
    wt/wt: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/wt | 38 | 36 | 38 | 112
    wt/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    wt/v | 13 | 16 | 17 | 46
    v/v: number analyzed (Participants) | 53 | 54 | 57 | 164
    v/v | 2 | 2 | 2 | 6
Menopause specific quality of life questionnaire mean score [Mean (Standard Deviation); unit: score on a scale] — MRS is a self-report questionnaire for evaluating the severity of menopausal symptoms in women, which contains 11 items. Each of the 11 symptoms contained a scoring scale from "0" (no complaints) to "4" (very severe symptoms). The total score will be calculated as the all items ranging from 0 to 44, with higher scores indicating worse symptoms. Population: The numbers are lower because there were no specimen available for analysis.
  score on a scale
    Vasomotor domain: number analyzed (Participants) | 48 | 54 | 57 | 159
    Vasomotor domain | 2.2 (1.9) | 2.5 (1.9) | 2.6 (1.9) | 2.4 (1.8)
    Psychosocial domain: number analyzed (Participants) | 48 | 54 | 57 | 159
    Psychosocial domain | 2.5 (1.3) | 2.3 (1.2) | 2.6 (1.5) | 2.5 (1.4)
    Physical domain: number analyzed (Participants) | 48 | 54 | 57 | 159
    Physical domain | 2.5 (1.1) | 2.3 (0.9) | 2.6 (1.4) | 2.5 (1.2)
    Sexual domain: number analyzed (Participants) | 48 | 54 | 57 | 159
    Sexual domain | 2.0 (1.4) | 1.9 (1.9) | 2.2 (1.8) | 2.1 (1.6)
    Overall: number analyzed (Participants) | 48 | 54 | 57 | 159
    Overall | 2.3 (0.9) | 2.2 (1.0) | 2.5 (1.1) | 2.4 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Time of Circulating Estradiol SPE in Each Arm
Description: LS means of percent change
Time Frame: baseline and 4-6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -89 [-95 to -83] | -85 [-98 to -73] | -60 [-78 to -42]

2. Secondary Outcome: Percent Change in Time of Circulating Estradiol LLE in Each Arm
Description: LS means of percent change
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -96 [-97 to -95] | -91 [-95 to -88] | -72 [-77 to -67]

3. Secondary Outcome: Percent Change of Circulating Estrone SPE
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 53 | 56 | 59
percent change | -93 [-98 to -88] | -89 [-96 to -83] | -73 [-81 to -52]

4. Secondary Outcome: Percent Change of Circulating Estrone LLE
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -99 [-99 to -98] | -96 [-97 to -93] | -78 [-85 to -62]

5. Secondary Outcome: Percent Change of Circulating Total Estrone
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -95 [-97 to -91] | -94 [-96 to -90] | -76 [-85 to -63]

6. Secondary Outcome: Percent Change of Circulating Estrone Sulfate
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -96 [-98 to -94] | -95 [-97 to -92] | -75 [-83 to -64]

7. Secondary Outcome: Percent Change of Circulating Androstenedione
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 59
percent change | 0 [-18 to 18] | 11 [-20 to 30] | 11 [-14 to 43]

8. Secondary Outcome: Percent Change of Circulating Testosterone
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 59
percent change | -19 [-33 to 0] | 0 [-25 to 0] | 0 [-20 to 18]

9. Secondary Outcome: Percent Change of Circulating Testosterone CLIA
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 53 | 56 | 60
percent change | 10 [-12 to 46] | 0 [-26 to 29] | 6 [-18 to 53]

10. Secondary Outcome: Percent Change of Circulating SHBG
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -29 [-36 to -17] | -15 [-23 to -7] | -5.5 [-17 to 1.2]

11. Secondary Outcome: Percent Change of Circulating Total Cholesterol
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 54 | 55 | 58
percent change | -4 [-17 to 4] | -5 [-9 to 5] | -1 [-9 to 6]

12. Secondary Outcome: Percent Change of Circulating HDL Cholesterol
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 54 | 56 | 58
percent change | -14 [-21 to -3] | -3 [-13 to 4] | -2 [-10 to 4]

13. Secondary Outcome: Percent Change of Circulating LDL Cholesterol
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 54 | 55 | 58
percent change | -1 [-18 to 13] | 0 [-13 to 10] | 0 [-13 to 9]

14. Secondary Outcome: Percent Change of Circulating Triglycerides
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 54 | 55 | 58
percent change | -7 [-22 to 25] | -1 [-19 to 17] | 5 [-17 to 23]

15. Secondary Outcome: Percent Change of Circulating Insulin
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | 3 [-15 to 46] | 9 [-19 to 47] | 4 [-22 to 33]

16. Secondary Outcome: Percent Change of Serum Glucose
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -1 [-7 to 9] | 1 [-9 to 9] | -2 [-5 to 6]

17. Secondary Outcome: Percent Change of HOMA IR
Description: Insulin Resistance Index (HOMA-IR) measures insulin resistance, calculated by fasting insulin (mU/L) multiplied by fasting glucose (mmol/L), and divided by a constant (22.5). A higher score indicates higher insulin resistance.
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 59
percent change | 8 [-18 to 55] | 15 [-19 to 53] | 6 [-26 to 39]

18. Secondary Outcome: Percent Change of Circulating Adiponectin
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -12 [-19 to 4] | -3 [-11 to 10] | -1 [-9 to 6]

19. Secondary Outcome: Percent Change of Circulating Leptin
Description: [(Final levels-baseline levels)/baseline levels]*100
Time Frame: baseline and 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 55 | 56 | 60
percent change | -16 [-33 to -3] | -5 [-22 to 8] | -4 [-17 to 20]

20. Secondary Outcome: Exemestane Blood Concentration at Surgery
Description: Final drug concentration
Time Frame: at surgery
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 54 | 55 | 58
pmol/L | 3217 [2320 to 4567] | 513 [341 to 727] | 24 [17 to 46]

21. Secondary Outcome: 17-OH Exemestane Blood Concentration at Surgery
Description: Final drug concentration
Time Frame: at surgery
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 54 | 55 | 58
pmol/L | 1069 [644 to 1657] | 196 [119 to 363] | 4 [4 to 22]

22. Secondary Outcome: Change of ER Expression (Cancer Tissue), Central Review
Description: Surgery level-biopsy level.
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: Abs change of % of positive tumor cells
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 50 | 53 | 55
Abs change of % of positive tumor cells | 0 [0 to 0] | 0 [-4 to 4] | 0 [0 to 0]

23. Secondary Outcome: Change of PgR Expression (Cancer Tissue), Central Review
Description: Surgery level-biopsy level.
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: Abs change of % of positive tumor cells
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 52 | 53 | 55
Abs change of % of positive tumor cells | -17 [-67 to -4] | -9 [-50 to 0] | -7 [-25 to 0]

24. Secondary Outcome: Change of Ki67% Expression (Cancer Tissue), Central Review
Description: Surgery level-biopsy level.
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: Abs change of % of positive tumor cells
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 52 | 53 | 55
Abs change of % of positive tumor cells | -7.5 [-11 to -3] | -5 [-10 to -1] | -4 [-8 to -1]

25. Secondary Outcome: Change of Ki67% Expression (Adjacent Non Cancer Tissue), Central Review
Description: Surgery level-biopsy level.
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: Absolute change of % of positive cells
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 28 | 22 | 27
Absolute change of % of positive cells | 0 [0 to 1] | 0 [-0.5 to 0.5] | 0 [-1 to 1]

26. Secondary Outcome: Estradiol Tissue Concentration at Surgery
Description: Final biomarker concentration
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: fmol/g wet weight
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 43 | 37 | 40
fmol/g wet weight
  cancer tissue | 15.5 [15.5 to 52.2] | 17.1 [15.5 to 125.3] | 128.8 [15.5 to 224.8]
  non cancer adjacent tissue | 15.5 [15.5 to 15.5] | 15.5 [15.5 to 15.5] | 15.5 [15.5 to 25.5]

27. Secondary Outcome: Estrone Tissue Concentration at Surgery
Description: Final biomarker concentration
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: fmol/g wet weight
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 43 | 37 | 40
fmol/g wet weight
  cancer tissue | 8.7 [4.5 to 21.7] | 28.1 [17.8 to 41.6] | 138.9 [53.2 to 246.7]
  non cancer adjacent tissue | 17.4 [4.8 to 33.0] | 37.8 [21.7 to 67.5] | 140.5 [68.2 to 233.3]

28. Secondary Outcome: Androstenedione Tissue Concentration at Surgery
Description: Final biomarker concentration.
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: fmol/g wet weight
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 43 | 37 | 40
fmol/g wet weight
  cancer tissue | 6864 [3324 to 8890] | 5314 [3692 to 6642] | 5564 [3194 to 8116]
  non cancer adjacent tissue | 10251 [6541 to 16103] | 12366 [8702 to 18654] | 10580 [5403 to 15003]

29. Secondary Outcome: Testosterone Tissue Concentration at Surgery
Description: Final biomarker concentration
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: fmol/g wet weight
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 43 | 37 | 40
fmol/g wet weight
  cancer tissue | 395 [273 to 567] | 396 [346 to 790] | 453 [314 to 700]
  non cancer adjacent tissue | 436 [273 to 654] | 464 [341 to 787] | 399 [299 to 570]

30. Secondary Outcome: Exemestane Tissue Concentration at Surgery
Description: Final drug concentration
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: fmol/g wet weight
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 43 | 37 | 40
fmol/g wet weight
  cancer tissue | 3807 [1663 to 7194] | 44 [44 to 291] | 44 [44 to 44]
  non cancer adjacent tissue | 17485 [6791 to 31985] | 435 [44 to 791] | 44 [44 to 44]

31. Secondary Outcome: 17 OH Exemestane Tissue Concentration at Surgery
Description: Final drug concentration
Time Frame: 4-6 weeks
Measure: Median (Inter-Quartile Range); unit: fmol/g wet weight
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 43 | 37 | 40
fmol/g wet weight
  cancer tissue | 338 [64 to 1360] | 65 [65 to 65] | 65 [65 to 65]
  non cancer adjacent tissue | 1343 [262 to 2758] | 65 [65 to 65] | 65 [65 to 65]

32. Secondary Outcome: Change in MenQoL Questionnaire Score
Description: MenQOL questionnaire assessed how bothered participants were with 31 symptoms. It contains domains: vasomotor (items 1-3); psychosocial (items 4-10); physical (items 11-26); sexual (items 27-29); in addition to nausea and indigestion. 31 individual symptoms are rated on a scale of 0 (not at all bothered) to 6 (extremely bothered). Total possible score ranged from 0 to 186. MenQOL summary score was calculated as mean of four domain scores (Physical function, Psychosocial function, Sexual function and Vasomotor function) ranging from 1 to 8, with higher scores indicating worse quality of life. Final score-baseline score
Time Frame: baseline and 4-6 weeks
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
Number analyzed (Participants) | 47 | 53 | 56
score on a scale
  Vasomotor domain | 0.41 (1.2) | 0.28 (1.4) | 0.51 (1.5)
  Psychosocial domain | -0.19 (0.98) | 0.06 (1.2) | -0.06 (1.1)
  Physical domain | -0.37 (0.77) | 0.07 (0.86) | -0.09 (0.67)
  Sexual domain | -0.45 (1.0) | -0.2 (1.7) | -0.52 (1.7)
  Overall | -0.15 (0.58) | 0.05 (0.79) | -0.06 (0.71)

33. Other Pre Specified Outcome: Proteomic Analysis
Description: The Proteomic Analysis was not performed.
Time Frame: 4-6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the first dose of exemestane through 30 days after the surgery
Arm/Group | Exemestane 25 mg QD | Exemestane 25 mg TIW | Exemestane 25 mg QW
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/57 | 0/57 | 0/62
Other Adverse Events (participants affected / at risk) | 36/57 | 40/57 | 37/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exemestane 25 mg QD (N=57) | Exemestane 25 mg TIW (N=57) | Exemestane 25 mg QW (N=62)
Bone Infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exemestane 25 mg QD (N=57) | Exemestane 25 mg TIW (N=57) | Exemestane 25 mg QW (N=62)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (8) | 11 (14) | 1 (1)
Fatigue (General disorders) | 3 (4) | 7 (9) | 3 (3)
Irritability (General disorders) | 1 (1) | 5 (5) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 2 (2)
GGT increased (Investigations) | 3 (3) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 2 (3) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 6 (8) | 8 (11) | 4 (6)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 3 (3) | 6 (6) | 7 (7)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 1 (1)
Hot Flashes (Vascular disorders) | 12 (12) | 11 (12) | 16 (16)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 (3) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT02598557/Prot_SAP_000.pdf